CLINICAL TRIAL: NCT04644991
Title: The Investigation of the Effect of Kinesiology Taping on Lumbar Region Structures and Balance in Transfemoral Amputees
Brief Title: The Effect of Kinesiology Taping on Lumbar Region Structures and Balance in Transfemoral Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20/100
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2020-11

CONDITIONS: Transfemoral Amputees; Kinesiology Taping
Keywords: amputation, transfemoral, thoracolumbal fascia, kinesiotape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Experimental): Experimental group consisting of transfemoral amputees who kinesiology tape will be applied
  Interventions: Other: Kinesiology taping; Other: Six minutes walking test
- ShamKinesiotape (Sham Comparator): The placebo group of transfemoral amputees who shame kinesiology tape will be applied
  Interventions: Other: Six minutes walking test; Other: Shame Kinesiology Tape

INTERVENTIONS:
Other: Kinesiology taping — Y-type kinesiology tape will be applied to the thoracolumbar fascia in experimental gruoup.
  Arms: Kinesiotape
Other: Six minutes walking test — Participants will be asked to walk as fast as they can for 6 minutes.
Other: Shame Kinesiology Tape — Sham kinesiology tape will be applied to the thoracolumbar fascia in sham gruoup.
  Arms: ShamKinesiotape

SUMMARY:
With the initiation of prosthesis use following lower extremity amputations, the body shows biomechanical changes according to the amputation level, and as a result, it develops adaptation mechanisms on both the healthy and ampute sides. It has been reported that the most common secondary pathology caused by these mechanisms developed to compensate the amputated side is lower back pain and adaptation mechanisms vary according to the presence of pain. Adaptation strategies in transfemoral amputees cause permanent changes in the connective tissue structure properties of the toracolumbar region and reduce the contribution of these structures to dynamic stability. It has been reported that with the fascia correction technique, one of the kinesiological taping techniques, the connective tissue fiber alignment can be rearranged and the degree of stiffness can be reduced. Before the intervention, biomechanical properties of the toracolumbar region structures with MyotonPro and postural stability measurements with TekScan will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-60
* Having unilateral transfemoral amputation
* Using prosthesis for at least 6 months
* Good prosthesis comfort

Exclusion Criteria:

* Body mass index>30
* Having a history of surgery in the lumbar region in past 6 months
* Participating in a physiotherapy and rehabilitation program for a low back pain past six months
* Neurological and / or orthopedic disorders other than amputation
* Having low back pain for at least 3 months before amputation

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Measurement of Postural Stability | Changes from baseline of center of gravity displacement at following 6 minutes walking test, at immediately after kinesiology tape applying and at 30. minutes following kinesiology tape applying.
  The center of gravity displacement (cm2) will be measured at standing position on force platform during 30sn
Measurement of Stiffness | Changes from baseline of stifness of thoracolumbal fascia at following 6 minutes walking test, at immediately after kinesiology tape applying and at 30. minutes following kinesiology tape applying.
  Stiffness of throcalumbar fascia will be measured using a myometer (MyotonPro, Myoton AS, Tallinn, Estonia).
Measurement of Creep | Changes from baseline of creep of thoracolumbal fascia at following 6 minutes walking test, at immediately after kinesiology tape applying and at 30. minutes following kinesiology tape applying
  Creep value of throcalumbar fascia will be measured using a myometer (MyotonPro, Myoton AS, Tallinn, Estonia).

SECONDARY OUTCOMES:
Low back pain | Changes from baseline of low back pain at following 6 minutes walking test, at immediately after kinesiology tape applying and at 30. minutes following kinesiology tape applying.
  Low back pain will be measured by Visual Analog Scale between 0 (no pain) and 10 (the most severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gailey R, Allen K, Castles J, Kucharik J, Roeder M. Review of secondary physical conditions associated with lower-limb amputation and long-term prosthesis use. J Rehabil Res Dev. 2008;45(1):15-29. doi: 10.1682/jrrd.2006.11.0147. PMID 18566923
- [Result] Morgenroth DC, Orendurff MS, Shakir A, Segal A, Shofer J, Czerniecki JM. The relationship between lumbar spine kinematics during gait and low-back pain in transfemoral amputees. Am J Phys Med Rehabil. 2010 Aug;89(8):635-43. doi: 10.1097/PHM.0b013e3181e71d90. PMID 20647781
- [Result] Murray AM, Gaffney BM, Davidson BS, Christiansen CL. Biomechanical compensations of the trunk and lower extremities during stepping tasks after unilateral transtibial amputation. Clin Biomech (Bristol). 2017 Nov;49:64-71. doi: 10.1016/j.clinbiomech.2017.08.010. Epub 2017 Aug 30. PMID 28888109
- [Result] Willard FH, Vleeming A, Schuenke MD, Danneels L, Schleip R. The thoracolumbar fascia: anatomy, function and clinical considerations. J Anat. 2012 Dec;221(6):507-36. doi: 10.1111/j.1469-7580.2012.01511.x. Epub 2012 May 27. PMID 22630613
- [Result] Yahia L, Rhalmi S, Newman N, Isler M. Sensory innervation of human thoracolumbar fascia. An immunohistochemical study. Acta Orthop Scand. 1992 Apr;63(2):195-7. doi: 10.3109/17453679209154822. PMID 1590057
- [Result] Stecco C, Day JA. The fascial manipulation technique and its biomechanical model: a guide to the human fascial system. Int J Ther Massage Bodywork. 2010 Mar 17;3(1):38-40. doi: 10.3822/ijtmb.v3i1.78. No abstract available. PMID 21589701
- [Result] Kalichman L, Vered E, Volchek L. Relieving symptoms of meralgia paresthetica using Kinesio taping: a pilot study. Arch Phys Med Rehabil. 2010 Jul;91(7):1137-9. doi: 10.1016/j.apmr.2010.03.013. PMID 20537313